CLINICAL TRIAL: NCT07351669
Title: The Performance of Spectral CT in Evaluating Treatment Response After Transarterial Chemoembolization for Hepatocellular Carcinoma: The SpecTRAIL Study
Brief Title: A Multicenter Prospective Study on the Performance of Spectral CT for Evaluating Treatment Response After TACE in Hepatocellular Carcinoma
Status: Not yet recruiting | Type: Observational
Sponsor: Zhongda Hospital (Other)
Responsible Party: Principal Investigator, Yuan-Cheng Wang, Head of Radiology, Zhongda Hospital
Other Study IDs: 2025ZDSYLL494-P01
Record Dates: First submitted 2025-12-29; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: HCC - Hepatocellular Carcinoma; TACE(Transcatheter Arterial Chemoembolization); CT
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
By comparing the diagnostic accuracy of spectral CT and conventional CT in evaluating treatment response efficacy after TACE, this study aims to investigate the diagnostic performance of spectral CT in assessing treatment response following TACE for hepatocellular carcinoma.

ELIGIBILITY:
Inclusion Criteria01:

1. Voluntary participation and ability to sign informed consent (post-TACE);
2. Age between 18 and 75 years;
3. Diagnosed as HCC based on pathology or clinical criteria, with a BCLC stage of A or B;
4. Patients undergo contrast-enhanced spectral CT 4-8 weeks after treatment and are assessed as complete response on conventional CT images;
5. Patients are scheduled to undergo surgical resection within one month, or DSA hepatic arteriography or contrast-enhanced MRI within one week. If none of these were planned, the patients were scheduled for imaging follow-up (CT or MRI) every 3 months (±15 days) for at least one year.

Inclusion Criteria02:

1. Voluntary participation and ability to sign informed consent (post-TACE, cTACE or DEB-TACE);
2. Age between 18 and 75 years;
3. Diagnosed as HCC based on pathology or clinical criteria, with a BCLC stage of A or B;
4. Patients plan to undergo liver tumor resection following TACE downstaging therapy;
5. Contrast-enhanced spectral CT was performed within 7 days before liver resection, after completion of TACE down-staging treatment.

Exclusion Criteria:

1. Contraindications to contrast-enhanced CT or contrast-enhanced MRI;
2. Presence of extrahepatic malignancies;
3. History of radiotherapy;
4. Poor image quality or incomplete clinical/imaging data; Withdrawal from the study midway.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients recruited from six comprehensive medical centers nationwide
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2026-01-20 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy of spectral CT in identifying nonviable HCC lesions. | From enrollment to the completion of the 1-year follow-up
  Two or more investigators independently evaluated the multiparametric spectral CT images of the patients using the mRECIST criteria. The imaging assessment results were recorded as CR, PR, PD, or SD. First, the agreement between spectral CT-based assessments and those obtained from conventional clinical CT was evaluated. Subsequently, the spectral CT imaging results were compared with the reference standard to assess the diagnostic accuracy of spectral CT.
Diagnostic Performance of Spectral CT for Residual Viable Hepatocellular Carcinoma After TACE. | From enrollment to the completion of the 1-year follow-up.
  Imaging Assessment Criteria:
  For target lesions, imaging evaluation was performed using the mRECIST and LI-RADS TRA v2024 criteria, with histopathological findings serving as the reference standard.
  Imaging Assessment Procedure:
  Two or more investigators independently and blindly reviewed the multiparametric spectral CT images of the patients. Lesions were assessed using the mRECIST criteria. The imaging assessment results were recorded as CR, PR, PD, or SD. The imaging findings were compared with the pathological reference standard to assess the diagnostic performance of spectral CT.